CLINICAL TRIAL: NCT01948882
Title: A Multi-Center, Multi-National Clinical Study to Evaluate the Safety and Effectiveness of the Essure® (Model ESS505) Device to Prevent Pregnancy in Women Who Are Seeking Permanent Contraception
Brief Title: Evaluation of Safety and Effectiveness of the Essure (Model ESS505) Device to Prevent Pregnancy in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 16973
Record Dates: First submitted 2013-09-19; First posted 2013-09-24 (Estimated); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Contraception
Keywords: Birth control

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- ESS505 (Experimental): All subjects that sign the informed consent and meet the eligibility criteria will be scheduled for an implant procedure.
  Interventions: Device: ESS505 (BAY1454033)

INTERVENTIONS:
Device: ESS505 (BAY1454033)

SUMMARY:
The Essure System is indicated for women who desire non-incisional permanent birth control (female sterilization) by occlusion of the fallopian tubes. The objective of the study is to evaluate the safety and effectiveness of the Essure System (Model ESS505) for permanent birth control in preventing pregnancy. The Essure ESS505 System includes a design modification that will be studied to determine if it provides immediate birth control, thereby removing the three months waiting period required for the commercially available Essure System Model 305 to be effective.

ELIGIBILITY:
Inclusion Criteria:

* Female, 21 to 44 years of age, inclusive
* Body weight within range of 90-300 lbs (40 - 136 kg)
* Sexually active (minimum of 4 coital acts per cycle)
* Willing to accept the risk of pregnancy while relying solely on the inserts for contraception
* Medical history indicates bilateral viable and patent fallopian tubes
* Agrees to fulfill local requirements for counseling and consent to contraception and sterilization, including any required waiting periods

Exclusion Criteria:

* Post-menopausal woman
* Suspected or confirmed pregnancy
* Post-partum or pregnancy termination ≤6 weeks of scheduled insert placement
* Past fallopian tube sterilization procedure and/or total or partial salpingectomies
* Diagnosis of any of the following: tubal, endometrial, or myometrial pathology (which may prevent fallopian tube ostia access), proximal tubal occlusion in either fallopian tube, unicornuate uterus, active or recent upper or lower pelvic infection, gynecologic malignancy
* Currently taking corticosteroids
* Known allergy to all contrast media available for use in hysterosalpingogram
* Scheduled to undergo concomitant intrauterine procedures at the time of insert placement (intrauterine device removal is not considered a concomitant procedure)
* Any general health condition or systemic disease that may represent, in the opinion of the physician, a potential increased risk associated with device use or pregnancy

Ages: 21 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 660 (Actual)
Dates: Start 2013-09-30 (Actual); Primary Completion 2015-09-16 (Actual); Study Completion 2024-09-12 (Actual)

PRIMARY OUTCOMES:
Number of confirmed pregnancies at 1 year among subjects told to rely on ESS505 for contraception | 1 year
  Evaluated after 6000 women-months of reliance have been accumulated
Reliance rate, defined as number of subjects told to rely on ESS505 after the Essure confirmation test divided by the number of subjects who had insert placement attempted | 3 months
  Evaluated after 3000 women-months of reliance have been accumulated (expected at the same time most subjects with implants have completed their 3 month follow-up visit)

SECONDARY OUTCOMES:
Number of confirmed pregnancies at 10 years among subjects told to rely on ESS505 for contraception | 10 years
Safety of the ESS505 placement procedure defined as number of subjects who experience an AE assessed as related to the ESS505 placement procedure divided by the number of subjects in who at least one ESS505 was introduced into the fallopian tube | On day of placement procedure
Safety of subsequent wearing of the insert defined as number of subjects who experience an AE assessed as related to wearing of ESS505 divided by the number of subjects in whom the presence of an AE could be assessed | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (22):
- United States (17):
  - Aurora, Colorado
  - Denver, Colorado
  - Wellington, Florida
  - Fort Wayne, Indiana
  - Newburgh, Indiana
  - Saginaw, Michigan
  - Rochester, Minnesota
  - New York, New York
  - The Bronx, New York
  - Asheville, North Carolina
  - Cincinnati, Ohio
  - Columbia, Ohio
  - Dallas, Texas
  - Houston, Texas
  - Irving, Texas
  - Norfolk, Virginia
  - Spokane, Washington
- Canada (2):
  - Hamilton, Ontario
  - Regina, Saskatchewan
- Zwolle, Netherlands
- Spain (2):
  - L'Hospitalet de Llobregat, Barcelona
  - Córdoba

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards — https://clinicaltrials.bayer.com/study/16973